CLINICAL TRIAL: NCT04554069
Title: Effect of Different Antihypertensive Treatment on Serum Uric Acid in Newly Diagnosed Hypertensive Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Mahran, Professor of Public Health and Community Medicine, Assiut University
Other Study IDs: Uric acid in Hypertension
Record Dates: First submitted 2020-09-05; First posted 2020-09-18 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of the influence of different antihypertensive drugs on serum uric acid in newly diagnosed hypertension patients.

DETAILED DESCRIPTION:
Hypertension is the most common condition seen in primary care and leads to myocardial infarction, stroke, renal failure, and death if not detected early and treated appropriately.

Thiazide-type diuretics, angiotensin-converting enzyme (ACE) inhibitors and some of angiotensin-II receptor blockers (ARB) were reported to reduce renal excretion of urate and increased serum uric acid levels, Beta-blockers also elevate serum uric acid levels.

Hyperuricemia is a risk factor for cardiovascular diseases. Hyperuricemia was found to correlate with hypertension excluding the influence of other factors such as age and renal function. Furthermore, many studies found that hyperuricemia was independently associated with cardiovascular events in patients treated with antihypertensive drugs.

It is important to control serum uric acid levels in hypertensive patients treated with antihypertensive drugs in order to reduce the risk of gout and cardiovascular events. There is a gap in knowledge in studies showing the effect of antihypertensive drugs on serum uric acid in newly diagnosed hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed hypertensive patients aged 30 years old and above will be invited to participate in this study

Exclusion Criteria:

1. Patients below 30 years old.
2. Patients with kidney disease.
3. Patients who are taking medications known to increase SUA as (Thiazide and Loop diuretics, Salicylates, Cyclosporin use) or decrease the level of uric acid in the urine as (Allopurinol, Febuoxstate).

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and Female participants aged 30 years old and above will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
The effect of different antihypertensive drugs on serum uric acid in newly diagnosed hypertension. | 6 months from baseline
  we will measure the change of the level of serum uric acid after 6 months from the treatment of antihypertensive durgs

SECONDARY OUTCOMES:
obesity | 6 months from baseline
  it will be measured by BMI (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Mahran, Professor, Principal Investigator — faculty of medicine

REFERENCES:
- [Background] Verdecchia P, Schillaci G, Reboldi G, Santeusanio F, Porcellati C, Brunetti P. Relation between serum uric acid and risk of cardiovascular disease in essential hypertension. The PIUMA study. Hypertension. 2000 Dec;36(6):1072-8. doi: 10.1161/01.hyp.36.6.1072. PMID 11116127
- [Background] Shankar A, Klein R, Klein BE, Nieto FJ. The association between serum uric acid level and long-term incidence of hypertension: Population-based cohort study. J Hum Hypertens. 2006 Dec;20(12):937-45. doi: 10.1038/sj.jhh.1002095. Epub 2006 Oct 5. PMID 17024135